CLINICAL TRIAL: NCT07079670
Title: A Phase 3 Open-Label, Single-Arm Study to Evaluate the Safety and Immunogenicity of an Omicron JN.1 Subvariant SARS-CoV-2 rS Vaccine Adjuvanted With Matrix-M
Brief Title: Safety and Immunogenicity of NVX-CoV2705
Acronym: COVID-19
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019nCoV-318
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Matrix-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NVX-CoV2705 (Experimental): NVX-CoV2705 vaccine in a 0.5 mL injection volume at an antigenic dose of 5 µg with 50 µg Matrix-M adjuvant.
  Interventions: Biological: NVX-CoV2705

INTERVENTIONS:
Biological: NVX-CoV2705 — Intramuscular (deltoid) injection at an antigenic dose of 5 µg with 50 µg Matrix-M adjuvant.
  Other Names: Omicron JN.1 Subvariant SARS-CoV-2 rS Vaccine Adjuvanted with Matrix-M

SUMMARY:
This study is a Phase 3 trial designed to check the safety and immune response to a new Omicron JN.1 COVID-19 vaccine. Study researchers will give a single dose of this vaccine, called NVX-CoV2705, to approximately 120 participants. This includes adults aged 65 and older, and individuals aged 12 to 64 who have existing health conditions that put them at high risk for severe COVID-19. All participants must have received a previous COVID-19 vaccine at least 90 days before joining this study. Study researchers will be closely monitoring participants for their immune response for 28 days and collecting safety data for 180 days after vaccination.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, single arm study to evaluate the safety and immunogenicity of a single dose of an Omicron JN.1 subvariant severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle vaccine (SARS-CoV-2 rS) adjuvanted with Matrix-M® (NVX-CoV2705) in participants ≥ 65 years of age and participants 12 through 64 years of age who have at least one underlying condition that puts them at high risk for severe outcomes from coronavirus disease 2019 (COVID 19) previously vaccinated with a COVID-19 vaccine ≥ 90 days prior to study vaccination. The goal will be to enroll a similar number of participants in the 2 age cohorts (≥ 65 years and 12 through 64 years) and in the 12 through 64 years age cohort, an effort will be made to enroll a similar number of participants in the 2 age subcohorts (12 through 17 years and 18 through 64 years).

Approximately 120 participants, approximately 60 participants in each age cohort and approximately 30 participants in each age subcohort, will be enrolled to receive a single dose of NVX-CoV2705 on Day 0 and remain on study for immunogenicity until Day 28 and safety data collection through 180 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, each individual must satisfy all the following criteria:

  1. Participants ≥ 65 years of age and participants 12 through 64 years who have at least one underlying condition that puts them at high risk of severe outcomes from COVID-19 at time of study vaccination. In each instance, the investigator's judgment may be exercised and other eligibility criteria must be respected.
  2. Previously vaccinated with a COVID-19 vaccine with the last dose administered ≥ 90 days prior to study vaccination (written or verbal confirmation by participant).
  3. Participant and parent(s)/caregiver(s) or legally acceptable representative willing and able to give informed consent and assent prior to study enrollment and to comply with study procedures.
  4. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to enrollment and through the end of the study.

     1. Condoms (male or female) with spermicide (if acceptable in country)
     2. Diaphragm with spermicide
     3. Cervical cap with spermicide
     4. Intrauterine device
     5. Oral or patch contraceptives
     6. Norplant®, Depo-Provera®, or other in country regulatory approved contraceptive method that is designed to protect against pregnancy
     7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle NOTE: Periodic abstinence (eg, calendar, ovulation, sympto-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  5. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and physical examination. Vital signs must be within medically acceptable ranges prior to study vaccination. If the individual has a diagnosis of hypertension, it must be stable and controlled with necessary medication.
  6. Agrees not to participate in any research involving receipt of investigational products (drug/biologic/device), including other SARS-CoV-2 prevention or treatment trials, for the duration of the study.

Exclusion Criteria:

* If an individual meets any of the following criteria, he or she is ineligible for this study:

  1. Current participation in research involving receipt of investigational products (drug/biologic/device).
  2. Received any other vaccine (except for a licensed seasonal influenza vaccine or rabies vaccine [if medically indicated]) within 28 days prior to study vaccination. For the influenza vaccine, a participant is eligible as long as the vaccine was administered ≥ 14 days prior to study vaccination.
  3. Any known history of allergies to products contained in the investigational product in the participant's lifetime.
  4. Any known history of anaphylaxis to any prior vaccine in the participant's lifetime.
  5. Known history of myocarditis or pericarditis in the participant's lifetime.
  6. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to study vaccination that, in the opinion of the investigator, might interfere with protocol compliance.
  7. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) that requires the use of immune modulators.

     NOTE: Stable endocrine disorders (eg, thyroiditis, pancreatitis), including stable diabetes mellitus with no history of diabetic ketoacidosis, are NOT excluded.
  8. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to study vaccination (Day 0).

     NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled or intranasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted.
  9. Received any prohibited medication (see Section 7.3), immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to study vaccination (Day 0).
  10. Active cancer (malignancy) on chemotherapy within 3 years prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
  11. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
  12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
  13. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).
  14. Temperature of > 38°C/≥ 100.4°F (oral measurement) or respiratory symptoms in the past 3 days (ie, cough, sore throat, difficulty breathing) leading up to Day 0.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-16 (Estimated); Primary Completion 2026-04-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Pseudovirus neutralization (ID50) of Omicron JN.1 subvariant vaccine expressed as GMFR | Day 28
  Pseudovirus neutralization (ID50) GMFR for the Omicron JN.1 subvariant at Day 28 following study vaccination.

SECONDARY OUTCOMES:
Pseudovirus neutralization (ID50) of Omicron JN.1 subvariant vaccine expressed as GMT | Day 28
  Pseudovirus neutralization (ID50) GMTs for the Omicron JN.1 subvariant at Day 28 following study vaccination.
Pseudovirus neutralization (ID50) of Omicron JN.1 subvariant vaccine expressed as SRR | Day 28
  SRRs in ID50 titers for the Omicron JN.1 subvariant assessed at Day 28 following study vaccination.
Number of Participants Reported Solicited Local and Systemic Adverse Events (AEs) | Day 28
  Number of participants reported solicited local and systemic adverse events (AEs)
Number of Participants Reported any unsolicited AEs and MAAEs | Day 28
  Incidence, severity, and relationship of any unsolicited AEs and MAAEs through 28 days after vaccination.
Number of Participants Reported MAAEs Attributed to Study Vaccine, Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs) | Day 180
  • Incidence and severity of treatment-related MAAEs, AESIs (predefined list, including PIMMCs and myocarditis and/or pericarditis), and SAEs through Day 180/EoS.